CLINICAL TRIAL: NCT03754894
Title: Effect of Using a Ready Made Plastic Stent With Apically Repositioned Flap in Augmentation of the Peri Implant Soft Tissue Randomized Clinical Study
Brief Title: Efficacy of a Ready Made Plastic Stent With Apically Repositioned Flap in Augmentation of the Peri Implant Soft Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, teaching assistant of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: per- 16 29 M
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Loss of Keratinized Gingiva Around Dental Implants
Keywords: dental implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- goup 1(with readymade plastic stent ) (Experimental): Will include 10 patients where combined full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement covered by ready-made plastic stent.
  Interventions: Device: ready made plastic stent application
- group 2 (control) (Experimental): Will include 10 patients where combined full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement then suturing the flap in place.
  Interventions: Procedure: simple interrupted sutures

INTERVENTIONS:
Device: ready made plastic stent application — full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement covered by ready-made plastic stent.
  Arms: goup 1(with readymade plastic stent )
Procedure: simple interrupted sutures — full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement and securing the flap with simple interrupted sutures
  Arms: group 2 (control)

SUMMARY:
Keratinized gingiva around dental implants are necessary to achieve esthetic appearance in the anterior teeth, also it is more resistant to abrasion, recession, less in plaque accumulation and inflammation, and easy to manipulate during stage two surgery and impression making in prosthetic stage. For the aforementioned reasons over year's authors have developed many techniques to increase the amount of keratinized gingiva around the dental implants such techniques are apically and laterally repositioned flaps , free gingival grafts, acellular dermal matrix allograft , coronally repositioned flap and sub epithelial connective tissue flaps . Huh et al compared the effects of the use of a ready-made plastic stent on the width of peri-implant keratinized mucosa with those of conventional methods. In addition, the effect of a plastic stent on peri-implant soft tissue was examined through histological observations. Reported that the width of the keratinized mucosa was significantly higher and the distance from the top of the implant platform to the mucogingival junction was significantly longer in the ready-made plastic stent group.

Thus this study will be performed to compare between the effect of the use of a ready- made plastic stent on the width of peri-implant keratinized tissue and that of conventional methods during first stage of implant surgery.

DETAILED DESCRIPTION:
This prospective clinical study will be conducted on Twenty patients will be selected from the outpatient clinic of Oral Medicine, Periodontology, and Oral Diagnosis department, Faculty of Dentistry, Ain Shams University This methodology will be reviewed by Ain shams university, faculty of dentistry research ethics committee

Inclusion criteria:

1. Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire.
2. Both genders.
3. Age from 20 -50 years old.
4. Having at least one missing tooth at Posterior area (premolars or molars).
5. Attached gingiva width below 3 mm.
6. Patient should agree to sign a written consent after the nature of the study will be explained.

Exclusion criteria:

1. Smokers ( >10 cigs/day ) .
2. Vulnerable groups (as pregnant females and decisional impaired individuals) will be excluded from the study.
3. Patients with poor oral hygiene or not willing to perform oral hygiene measures.
4. Prisoners and handicapped patients.
5. Patients with periodontal or periapical infections.

Patients met the eligibility criteria will be randomly allocated using computer assisted randomization through numbered sealed envelopes into two treatment modalities groups: -

Group I (with ready-made plastic stent): Will include 10 patients where combined full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement covered by ready-made plastic stent.

Group II (control): Will include 10 patients where combined full / partial thickness apically repositioned flap with paracrestal lingual incision will be performed for implant placement followed by healing abutment placement then suturing the flap in place.

All patients will receive healing abutments in first stage of implant surgery.

This proposal will be reviewed by the research ethics committee, the procedure will be fully explained to the patients and they will sign an informed consent

ELIGIBILITY:
Inclusion Criteria:

- 1- Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire.

2- Both genders. 3- Age from 20 -50 years old. 4- Having at least one missing tooth at Posterior area (premolars or molars). 5- Attached gingiva width below 3 mm. 6- Patient should agree to sign a written consent after the nature of the study will be explained.

Exclusion Criteria:

1. Smokers ( >10 cigs/day ) .(Ata-Ali et al , 2015)
2. Vulnerable groups (as pregnant females and decisional impaired individuals) will be excluded from the study.
3. Patients with poor oral hygiene or not willing to perform oral hygiene measures.
4. Prisoners and handicapped patients.
5. Patients with periodontal or periapical infections.

   -

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
increasing attached gingiva width around implant | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams Dental School, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamdy A, Abd El Gaber HK, Ghalwash DM, Abbas WM. Effect of Using a Plastic Stent with Apically Repositioned Flap in Peri-Implant Soft Tissue Augmentation: A Randomized Controlled Clinical Trial. Int J Dent. 2021 May 18;2021:5590400. doi: 10.1155/2021/5590400. eCollection 2021. PMID 34113381